CLINICAL TRIAL: NCT07057908
Title: A Prospective Observational Study Comparing Tracheal Intubation Via Video Laryngeal Mask Airway and Video Laryngoscope in Adult Patients Undergoing Elective Surgery
Brief Title: Comparison of Intubation Using Video Laryngeal Mask and Video Laryngoscope in Elective Surgical Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/10/1
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Airway Management; Tracheal Intubation; Elective Surgeries; Videolaryngoscopy; Anaesthesia
Keywords: Video Laryngoscope; Video Laryngeal Mask Airway; SaCoVLM; Intubation Success Rate; Observational Study; Elective Surgical Patients
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video Laryngoscope: Tracheal intubation using a video laryngoscope assisted with a bougie in adult patients undergoing elective surgery.
  Interventions: Procedure: Video Laryngeal Mask Airway (SaCoVLM) Intubation with Bougie
- Video Laryngeal Mask Airway (SaCoVLM): Tracheal intubation performed through a video laryngeal mask airway (SaCoVLM) with bougie assistance in adult patients undergoing elective surgery.
  Interventions: Procedure: Video Laryngoscope Intubation with Bougie

INTERVENTIONS:
Procedure: Video Laryngoscope Intubation with Bougie — Participants in this group will undergo tracheal intubation using a video laryngoscope under general anesthesia. After induction, a standard bougie will be advanced through the vocal cords under video guidance, and the endotracheal tube will be railroaded over the bougie into the trachea.
  The primary outcome will be intubation time, measured from insertion of the device until confirmation of successful tracheal intubation. Additional parameters such as intubation success rate, ease of insertion, and complications (e.g., desaturation, airway trauma, failed attempts) will also be recorded. No extra procedures will be performed beyond routine airway management.
  Groups: Video Laryngeal Mask Airway (SaCoVLM)
Procedure: Video Laryngeal Mask Airway (SaCoVLM) Intubation with Bougie — Participants in this group will undergo tracheal intubation using a video laryngeal mask airway (SaCoVLM) under general anesthesia. After successful placement of the device, a standard bougie will be inserted through the SaCoVLM's dedicated lumen, and an endotracheal tube will be advanced over the bougie into the trachea under video guidance.
  The primary outcome will be intubation time, defined as the duration from device insertion to confirmation of successful intubation. Secondary outcomes include intubation success rate, ease of insertion, and complications such as desaturation, trauma, or failed attempts. As both techniques are part of routine practice, no additional risks will be introduced.
  Groups: Video Laryngoscope

SUMMARY:
This study compares two airway devices that are commonly used during elective surgery: the video laryngeal mask airway (VLM) and the video laryngoscope (VLS). Both are part of routine anesthesia practice. Our main focus is to measure how long intubation takes with each device and to see how successful the intubation is. The study does not involve any extra procedures or risks; everything will be carried out as part of normal patient care.

DETAILED DESCRIPTION:
In this prospective observational study, we will compare two airway devices commonly used during elective surgeries: the video laryngeal mask airway (SaCoVLM) and the video laryngoscope. The study will involve adult patients (18 years and older, ASA physical status I-III) scheduled to undergo surgery under general anesthesia at Samsun University Training and Research Hospital.

Patients will be assigned to one of two groups. In one group, intubation will be performed using a video laryngoscope; in the other group, a video laryngeal mask will be used. In both groups, tracheal intubation will be carried out with the assistance of a bougie after device placement.

The primary outcome of the study will be intubation time, defined as the duration from insertion of the device until successful confirmation of tracheal intubation. Secondary outcomes will include ease of insertion, the need for additional maneuvers, and complications such as desaturation, trauma, or failed attempts.

Since both techniques, as well as bougie use, are already part of routine anesthesia practice, no extra interventions or risks will be introduced. The aim of the study is to compare the performance of these two devices under everyday clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Patients scheduled for elective surgical procedures
* Patients classified as ASA Physical Status I-III
* Patients undergoing general anesthesia

Exclusion Criteria:

* Patients younger than 18 years
* Patients undergoing emergency surgery
* Patients with difficult airway predictors, such as:

Mallampati score ≥ 3

Thyromental distance < 6 cm

Mouth opening < 3 cm

* Patients with anatomical abnormalities or surgical history involving the oropharynx, larynx, or airway
* Patients with conditions contraindicating head or neck manipulation (e.g., cervical instability, upper airway tumors)

Pregnant patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older, classified as ASA I to III, who are scheduled to undergo elective surgical procedures under general anesthesia. All participants will require tracheal intubation using either a video laryngoscope or a video laryngeal mask airway (SaCoVLM), both with bougie assistance.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Time to Successful Intubation | Intraoperative (from tube passing the upper incisors to the third ETCO₂ waveform)
  The time from when the endotracheal tube passes the upper incisors to the appearance of three consecutive end-tidal CO₂ (ETCO₂) waveforms on the capnograph. This will be used as the objective marker of successful tracheal intubation. Timing will be recorded in seconds by an independent observer using a stopwatch.

SECONDARY OUTCOMES:
First-Attempt Intubation Success Rate | Immediately after intubation
  Defined as successful tracheal intubation on the first attempt, confirmed by visualization of three consecutive ETCO₂ waveforms and bilateral chest expansion.
  The outcome will be recorded as a binary variable:
  Yes = Successful on first attempt
  No = Failed or required multiple attempts
Insertion-Related Complications | Intraoperative and early postoperative period (0-30 minutes)
  Complications related to the airway device or bougie use, including desaturation (SpO₂ < 92%), oropharyngeal trauma (visible bleeding), or need for additional maneuvers.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice S Kuşderci, Study Director — Samsun University Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sargin M, Uluer MS. Comparison of McGrath((R)) Series 5 video laryngoscope with Macintosh laryngoscope: A prospective, randomised trial in patients with normal airways. Pak J Med Sci. 2016 Jul-Aug;32(4):869-74. doi: 10.12669/pjms.324.10037. PMID 27648030
- [Background] Levitan RM, Ochroch EA, Kush S, Shofer FS, Hollander JE. Assessment of airway visualization: validation of the percentage of glottic opening (POGO) scale. Acad Emerg Med. 1998 Sep;5(9):919-23. doi: 10.1111/j.1553-2712.1998.tb02823.x. PMID 9754506
- [Background] Sun Y, Huang L, Xu L, Zhang M, Guo Y, Wang Y. The Application of a SaCoVLMTM Visual Intubation Laryngeal Mask for the Management of Difficult Airways in Morbidly Obese Patients: Case Report. Front Med (Lausanne). 2021 Nov 18;8:763103. doi: 10.3389/fmed.2021.763103. eCollection 2021. PMID 34869469